CLINICAL TRIAL: NCT03613545
Title: Efficacy and Safety of Fecal Microbiota Transplantation for Irritable Bowel Syndrome
Brief Title: Fecal Microbiota Transplantation for Irritable Bowel Syndrome
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Guangzhou First People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: K-2017-078-02
Record Dates: First submitted 2018-07-27; First posted 2018-08-03 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-07

CONDITIONS: Irritable Bowel Syndrome; Fecal Microbiota Transplantation
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Fecal Microbiota Transplantation; Probiotics; Anti-Bacterial Agents; Antidepressive Agents; Rifaximin

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant
Masking Description: Masking only Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- fecal microbiota transplantation (Experimental): fecal microbiota transplantation
  Interventions: Procedure: fecal microbiota transplantation
- placebo fecal microbiota transplantation (Sham Comparator): Infusion of sham
  Interventions: Procedure: Infusion of sham
- Traditional treatments (Sham Comparator): Traditional treatments according to associated guidelines such as probiotics, antibiotics or antidepressants
  Interventions: Drug: probiotics, antibiotics or antidepressants

INTERVENTIONS:
Procedure: fecal microbiota transplantation — 200 mL of prepared fecal microbiota suspension from heathy donors' fresh feces was injected into the colon
  Arms: fecal microbiota transplantation
Procedure: Infusion of sham — Infusion of sham
  Arms: placebo fecal microbiota transplantation
Drug: probiotics, antibiotics or antidepressants — Drugs such as probiotics, antibiotics, antidepressants
  Other Names: rifaximin; Clostridium butyricum TO-A
  Arms: Traditional treatments

SUMMARY:
Fecal microbiota transplantation (FMT) is a strategy that infuses a fecal suspension containing a healthy donor's microbiota into a patient's gut to restore his/her intestinal microbiome. FMT has a higher cure rate than standard antibiotic treatment for recurrent Clostridium difficile infections,and shows promising results in Inflammatory bowel disease（IBD）.However, few studies have evaluated whether FMT is effective to treat Irritable bowel syndrome(IBS).The investigators propose to determine the efficiency and safety of FMT in patients with Irritable bowel syndrome.

DETAILED DESCRIPTION:
The present clinical trial aims to re-establish a gut functionality state of intestinal flora through FMT as a therapy for Irritable bowel syndrome(IBS). We established a standard microbiota isolation from donated fresh stool in lab. Then the microbiota is transplanted to the whole colon through a tube. Patients from Guangzhou First People's Hospital in this study will be assigned to receive FMT at least two times according to associated guidelines and follow-up for at least six months. Questionnaires will be used to assess participants at study start and at study completion.

ELIGIBILITY:
Inclusion Criteria:

To be considered eligible for enrolment into the study, subjects must:

* Be able to give written informed consent.
* Males and females aged >18 and <75
* Have IBS as defined by the Rome IV criteria

Exclusion Criteria:

Subjects will be excluded from the study if they meet any of the below criteria:

* pregnant or having a follow-up of less than 6 months;
* unable to give informed consent;
* suffering from other severe disease ,including liver and kidney failure, cancers, intestinal diseases, inflammatory bowel disease, C difficile infection;
* unable to undergo endoscopy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-08-10 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Irritable Bowel Syndrome assessed by Symptom Severity Score (IBS-SSS) | baseline; one month;three months;six months
  This questionnaire was used for assessing IBS severity. Scores of five questions were calculated with the Visual Analogue Scale (VAS) scale: the severity of abdominal pain, the frequency of abdominal pain, the severity of abdominal distention, dissatisfaction with bowel habits and interference with quality of life. The scores ranged from 0 to 500, a higher score indicating worse condition :<75 indicated remission; 75-175 indicated mild IBS;176-300 indicated moderate IBS; and > 300 indicated severe IBS .

SECONDARY OUTCOMES:
Change in Irritable Bowel Syndrome assessed by Quality of Life (IBS-QOL) Questionnaire Scores | baseline; one month;three months;six months
  The IBS-QOL questionnaire consisted of 34 items, covering eight aspects (dysphoria, interference with activity, body image, health worry, food avoidance,social reaction, sexual dysfunction, and relationships). Each item was rated on a 5-point Likert scale(1 = not at all, 5 = a great deal). Total scores were transformed to a 0±100 scale ranging from 0 (maximum quality of life) to 100 (poor quality of life).
Change in Depression and Anxiety assessed by Hamilton Depression Rating Scale (HAMD) and Hamilton Anxiety Rating Scale(HAMA) | baseline; one month;three months;six months
  The Hamilton Depression Rating Scale (HAMD) and Hamilton Anxiety Rating Scale (HAMA) were used to evaluate the mental and psychological states of patients. HAMD scores were graded as follows: 8-19, mild depression; 20-34, moderate depression; ≥35, severely depression. HAMA scores were graded as follows: 14-20, mild anxiety; 21-28, moderate anxiety;≥29 , severe anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Hongli Huang, MM, Principal Investigator — Guangzhou First People's Hospital
Locations (1):
- Guangzhou First People's Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Distrutti E, Monaldi L, Ricci P, Fiorucci S. Gut microbiota role in irritable bowel syndrome: New therapeutic strategies. World J Gastroenterol. 2016 Feb 21;22(7):2219-41. doi: 10.3748/wjg.v22.i7.2219. PMID 26900286